CLINICAL TRIAL: NCT02266017
Title: An Accessible Mobile Health Behavioral Intervention For Cancer Pain
Brief Title: Mobile Pain Coping Skills Training for Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00054792; Research Scholars Grant (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2014-09-02; First posted 2014-10-16 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Mobile Pain Coping Skills Training; In Person Pain Coping Skills Training
Keywords: pain; coping; mhealth; cancer
MeSH Terms: conditions — Pain; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile Pain Coping Skills Training (Experimental): Coping Skills Training for pain will be delivered to participants using video-conferencing via a tablet computer.
  Interventions: Behavioral: Pain Coping Skills Training
- In person Pain Coping Skills Training (Active Comparator): Participants will be provided with an in-person pain coping skills training intervention
  Interventions: Behavioral: Pain Coping Skills Training

INTERVENTIONS:
Behavioral: Pain Coping Skills Training

SUMMARY:
Pain in cancer patients is estimated to be as high as 90% and results in physical and psychological disability. Behavioral interventions that increase patients' confidence in their ability to manage their pain have been shown to be beneficial. Behavioral interventions for cancer pain teach patients how their thoughts and feelings can influence their pain and specific strategies (e.g., relaxation) for decreasing cancer pain. However, despite guidelines recommending such interventions be used in the care of cancer patients with pain, they are not routinely used. A critical barrier to the use of behavioral interventions is that patients have difficulties attending appointments which are typically offered at the medical center during normal business hours. Mobile health (mHealth) technologies provide new opportunities to decrease such barriers. The investigators have developed a new mHealth approach that may increase the use of behavioral cancer pain interventions and ultimately lead to greater use of interventions that can decrease pain and disability.

The investigators propose to test an approach that uses mHealth technologies to deliver a behavioral cancer pain intervention to patients in their home using a tablet computer (e.g., iPad) and video-conferencing (e.g., Skype). The investigators will randomly assign 160 cancer patients with breast, lung, prostate, or colorectal cancer pain to receive either mHealth Pain Coping Skills Training system (mPCST) or to receive a traditional in-person pain coping skills training intervention protocol (PCST-trad) at the medical center. The investigators will test whether the mPCST is more accessible to patients than PCST-trad. The investigators expect that mPCST, compared to PCST-trad, will: a) be more feasible meaning that more patients will complete it in a timely manner; b) create less burden meaning it is easier for patients physically, emotionally, and financially to participate; c) increase engagement meaning that patients will practice skills more and have more understanding of the material; and d) be more overall acceptable to patients. the investigators also expect that patients who find this intervention more feasible, less burdensome, more engaging, and more acceptable will be more likely to experience decreased pain, physical disability, and psychological disability, and increased confidence in their ability to manage their pain.

The investigators' goal is to use mHealth technologies to facilitate wide-spread use of behavioral cancer pain interventions. Increased use of mHealth behavioral cancer pain interventions will particularly benefit patients living far from medical centers (e.g., rural), experiencing cancer-related physical challenges, and facing other practical barriers (e.g., transportation, work) to in-person interventions. These outcomes could lead to future work evidencing that mHealth behavioral interventions could be applied to other areas of quality of life in cancer patients (e.g., fatigue) and/or in other samples of patients with persistent pain (e.g., arthritis).

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of 6 or more months
* Clinical pain rating of 3/10
* Primary diagnosis of breast, lung, prostate, or colorectal cancer in last year

Exclusion Criteria:

* Cognitive impairment
* Metastases to brain
* Treatment for serious psychological disorder in last 6 months
* Current or past engagement in pain coping skills training for cancer pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Change in Pain | Pre Study Intervention, Post Study Intervention & 3-month follow-up after post intervention
  Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Tamara J Somers, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States